CLINICAL TRIAL: NCT02966145
Title: The Four-Repeat Tauopathy Neuroimaging Initiative
Brief Title: 4-Repeat Tauopathy Neuroimaging Initiative - Cycle 2
Acronym: 4RTNI-2
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4RTNI-2; 2R01AG038791-06A1 (NIH)
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Corticobasal Degeneration (CBD); Corticobasal Syndrome (CBS); Cortical-basal Ganglionic Degeneration (CBGD); Progressive Supranuclear Palsy (PSP); Nonfluent Variant Primary Progressive Aphasia (nfvPPA); Oligosymptomatic/Variant Progressive Supranuclear Palsy (o/vPSP)
Keywords: CBD; CBS; CBGD; PSP; nfvPPA; oPSP; vPSP; o/vPSP; Corticobasal Degeneration; Corticobasal Syndrome; Cortocal-basal Ganglionic Degeneration; Progressive Supranuclear Palsy; Nonfluent Variant Primary Progressive Aphasia; Oligosymptomatic Progressive Supranuclear Palsy; Variant Progressive Supranuclear Palsy; Biomarker; Neuroimaging; MRI; PET; Tau; Oculomotor; Retinal Imaging
MeSH Terms: conditions — Corticobasal Degeneration; Supranuclear Palsy, Progressive; Pick Disease of the Brain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, cell lines and cerebrospinal fluid (CSF) will be retained by study investigators and stored at NIH-funded repositories.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PSP & CBD: Observational study of participants with a diagnosis of Progressive Supranuclear Palsy or Corticobasal Degeneration (also called Corticobasal Syndrome or Cortical-basal Ganglionic Degeneration).
  Interventions: Other: Observational Study
- o/vPSP: Observational study of participants with a diagnosis of an oligosymptomatic or variant Progressive Supranuclear Palsy syndrome.
  Interventions: Other: Observational Study
- Normal Volunteers: Observational study of participants with no known diagnosis of a neurological or neurodegenerative condition, and no known history of memory complaints.
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study

SUMMARY:
The goal of this study is to identify the most reliable methods of analysis for tracking CBD, PSP, and o/vPSP over time. The results from this study may be used in the future to calculate statistical power for clinical drug trials. The study will also provide information about the relative value of novel imaging techniques for diagnosis, as well as the value of imaging techniques versus testing of blood, urine, and cerebrospinal fluid (CSF) 'biomarkers'.

ELIGIBILITY:
Inclusion Criteria:

* No known history of neurological disease, or meet criteria for one of the following: Corticobasal Syndrome or Degeneration (CBS or CBD); Progressive Supranuclear Palsy (PSP); or Oligo- or Variant- Progressive Supranuclear Palsy (o/vPSP)
* Needs a reliable study partner who has frequent contact with the participant, who is available to provide information about the participant, and who can accompany the participant to research visits as needed
* Must be willing and able to undergo testing procedures, which include longitudinal follow-up visits
* Must be able to walk five steps with minimal assistance

Exclusion Criteria:

* Significant neurological disease other than CBD, PSP, or a variant PSP syndrome.
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, or metal fragments or metal objects in the eyes, skin, or body
* In the site investigator's opinion, inability to complete sufficient key study procedures, or some other equivalent assessment of impairment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with Corticobasal Syndrome (CBS), Corticobasal Degeneration (CBD), Progressive Supranuclear Palsy, or Oligo- or Variant- Progressive Supranuclear Palsy (o/vPSP); Healthy Volunteers.
Sampling Method: Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2016-01; Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Tau-PET Brain Scan | Baseline, 1-year, and 2-years.
  Change from Baseline of Tau protein distribution in the brain.
Amyloid-PET Brain Scan | Baseline
  Presence of Amyloid in the brain at Baseline.
Brain Volume on MRI | Baseline, 6-months, 1-year, and 2-years.
  Change from Baseline of brain tissue volume.
Progressive Supranuclear Palsy Rating Scale (PSPRS) | Baseline, 6-months, 1-year, and 2-years.
  Change from Baseline of this rating scale.
Corticobasal Degeneration Functional Scale (CBDFS) | Baseline, 6-months, 1-year, and 2-years.
  Change from Baseline of this rating scale.
Eye Movement Function | Baseline, 6-months, 1-year, and 2-years.
  Change from Baseline of eye movement function.
Retinal Imaging | Baseline, 6-months, 1-year, and 2-years.
  Change from Baseline of retinal thickness.
UDS Neuropsychological Testing Battery, including supplemental FTLD Module | Baseline, 6-months, 1-year, and 2-years.
  Change fromm Baseline of cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Adam L Boxer, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (8):
- United States (7):
  - University of California, San Diego (UCSD), San Diego, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - Harvard University - Massachusetts General Hospital, Charlestown, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data are available by request .

REFERENCES:
- [Background] Armstrong MJ, Litvan I, Lang AE, Bak TH, Bhatia KP, Borroni B, Boxer AL, Dickson DW, Grossman M, Hallett M, Josephs KA, Kertesz A, Lee SE, Miller BL, Reich SG, Riley DE, Tolosa E, Troster AI, Vidailhet M, Weiner WJ. Criteria for the diagnosis of corticobasal degeneration. Neurology. 2013 Jan 29;80(5):496-503. doi: 10.1212/WNL.0b013e31827f0fd1. PMID 23359374
- [Background] Boxer AL, Lang AE, Grossman M, Knopman DS, Miller BL, Schneider LS, Doody RS, Lees A, Golbe LI, Williams DR, Corvol JC, Ludolph A, Burn D, Lorenzl S, Litvan I, Roberson ED, Hoglinger GU, Koestler M, Jack CR Jr, Van Deerlin V, Randolph C, Lobach IV, Heuer HW, Gozes I, Parker L, Whitaker S, Hirman J, Stewart AJ, Gold M, Morimoto BH; AL-108-231 Investigators. Davunetide in patients with progressive supranuclear palsy: a randomised, double-blind, placebo-controlled phase 2/3 trial. Lancet Neurol. 2014 Jul;13(7):676-85. doi: 10.1016/S1474-4422(14)70088-2. Epub 2014 May 27. PMID 24873720
- [Background] Fagan AM, Shaw LM, Xiong C, Vanderstichele H, Mintun MA, Trojanowski JQ, Coart E, Morris JC, Holtzman DM. Comparison of analytical platforms for cerebrospinal fluid measures of beta-amyloid 1-42, total tau, and p-tau181 for identifying Alzheimer disease amyloid plaque pathology. Arch Neurol. 2011 Sep;68(9):1137-44. doi: 10.1001/archneurol.2011.105. Epub 2011 May 9. PMID 21555603
- [Background] Golbe LI, Ohman-Strickland PA. A clinical rating scale for progressive supranuclear palsy. Brain. 2007 Jun;130(Pt 6):1552-65. doi: 10.1093/brain/awm032. Epub 2007 Apr 2. PMID 17405767
- [Background] Heuer HW, Mirsky JB, Kong EL, Dickerson BC, Miller BL, Kramer JH, Boxer AL. Antisaccade task reflects cortical involvement in mild cognitive impairment. Neurology. 2013 Oct 1;81(14):1235-43. doi: 10.1212/WNL.0b013e3182a6cbfe. Epub 2013 Aug 28. PMID 23986300
- [Background] Litvan I, Agid Y, Calne D, Campbell G, Dubois B, Duvoisin RC, Goetz CG, Golbe LI, Grafman J, Growdon JH, Hallett M, Jankovic J, Quinn NP, Tolosa E, Zee DS. Clinical research criteria for the diagnosis of progressive supranuclear palsy (Steele-Richardson-Olszewski syndrome): report of the NINDS-SPSP international workshop. Neurology. 1996 Jul;47(1):1-9. doi: 10.1212/wnl.47.1.1. PMID 8710059
- [Background] Scherling CS, Hall T, Berisha F, Klepac K, Karydas A, Coppola G, Kramer JH, Rabinovici G, Ahlijanian M, Miller BL, Seeley W, Grinberg LT, Rosen H, Meredith J Jr, Boxer AL. Cerebrospinal fluid neurofilament concentration reflects disease severity in frontotemporal degeneration. Ann Neurol. 2014 Jan;75(1):116-26. doi: 10.1002/ana.24052. Epub 2014 Jan 2. PMID 24242746
- [Background] Stamelou M, de Silva R, Arias-Carrion O, Boura E, Hollerhage M, Oertel WH, Muller U, Hoglinger GU. Rational therapeutic approaches to progressive supranuclear palsy. Brain. 2010 Jun;133(Pt 6):1578-90. doi: 10.1093/brain/awq115. Epub 2010 May 14. PMID 20472654
- [Background] Steele JC, Richardson JC, Olszewski J. Progressive supranuclear palsy: a heterogeneous degeneration involving the brain stem, Basal Ganglia and cerebellum with vertical gaze and pseudobulbar palsy, nuchal dystonia and dementia. Semin Neurol. 2014 Apr;34(2):129-50. doi: 10.1055/s-0034-1377058. Epub 2014 Jun 25. No abstract available. PMID 24963673
- [Background] Wagshal D, Sankaranarayanan S, Guss V, Hall T, Berisha F, Lobach I, Karydas A, Voltarelli L, Scherling C, Heuer H, Tartaglia MC, Miller Z, Coppola G, Ahlijanian M, Soares H, Kramer JH, Rabinovici GD, Rosen HJ, Miller BL, Meredith J, Boxer AL. Divergent CSF tau alterations in two common tauopathies: Alzheimer's disease and progressive supranuclear palsy. J Neurol Neurosurg Psychiatry. 2015 Mar;86(3):244-50. doi: 10.1136/jnnp-2014-308004. Epub 2014 Jun 4. PMID 24899730
- [Background] Scotton WJ, Shand C, Todd EG, Bocchetta M, Kobylecki C, Cash DM, VandeVrede L, Heuer HW, Quaegebeur A, Young AL, Oxtoby N, Alexander D, Rowe JB, Morris HR; PROSPECT Consortium; Boxer AL; 4RTNI Consortium; Rohrer JD, Wijeratne PA. Distinct spatiotemporal atrophy patterns in corticobasal syndrome are associated with different underlying pathologies. Brain Commun. 2025 Feb 11;7(2):fcaf066. doi: 10.1093/braincomms/fcaf066. eCollection 2025. PMID 40070441
- [Result] Wise A, Li J, Yamakawa M, Loureiro J, Peterson B, Worringer K, Sivasankaran R, Palma JA, Mitic L, Heuer HW, Lario-Lago A, Staffaroni AM, Clark A, Taylor J, Ljubenkov PA, Vandevrede L, Grinberg LT, Spina S, Seeley WW, Miller BL, Boeve BF, Dickerson BC, Grossman M, Litvan I, Pantelyat A, Tartaglia MC, Zhang Z, Wills AA, Rexach J, Rojas JC, Boxer AL; as the 4-Repeat Tauopathy Neuroimaging Initiative. CSF Proteomics in Patients With Progressive Supranuclear Palsy. Neurology. 2024 Aug 13;103(3):e209585. doi: 10.1212/WNL.0000000000209585. Epub 2024 Jul 3. PMID 38959435
- [Result] Garcia-Cordero I, Anastassiadis C, Khoja A, Morales-Rivero A, Thapa S, Vasilevskaya A, Davenport C, Sumra V, Couto B, Multani N, Taghdiri F, Anor C, Misquitta K, Vandevrede L, Heuer H, Tang-Wai D, Dickerson B, Pantelyat A, Litvan I, Boeve B, Rojas JC, Ljubenkov P, Huey E, Fox S, Kovacs GG, Boxer A, Lang A, Tartaglia MC; 4-R-Tauopathy Neuroimaging Initiative Consortium, and the Alzheimer's Disease Neuroimaging Initiative. Evaluating the Effect of Alzheimer's Disease-Related Biomarker Change in Corticobasal Syndrome and Progressive Supranuclear Palsy. Ann Neurol. 2024 Jul;96(1):99-109. doi: 10.1002/ana.26930. Epub 2024 Apr 5. PMID 38578117